CLINICAL TRIAL: NCT06684366
Title: Chronic Coronary Syndrome...real Practice and Guidelines...A Single Center Registery
Brief Title: Chronic Coronary Syndrome Real Practice and Guidelines
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samar Mohamed Gad Bayoumi, residuent doctor, Assiut University
Other Study IDs: Chronic coronary Syndrome
Record Dates: First submitted 2024-10-24; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: chronic coronary syndrome
MeSH Terms: interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Simvastatin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Statins (atorvastatin or simvastatin) — A resting transthoracic echocardiogram Non-invasive functional imaging for myocardial ischemia or coronary computed tomography angiography (CCTA) is recommended as the initial test for diagnosing CAD in symptomatic patients in whom obstructive CAD cannot be excluded by clinical assessment alone

SUMMARY:
Evaluate Adherence to the 2019 ESC Guidelines and standard care protocols for managing patients with the chronic coronary syndrome within the center

DETAILED DESCRIPTION:
Coronary artery disease (CAD) refers to the presence of atherosclerotic plaques in the coronary arteries, Which can be non-obstructive or obstructive. It represents a major cause of morbidity, mortality, Hospitalization and health expenditure.

The most recent European Guidelines for the diagnosis and management of CCS delineate six common CCS scenarios: patients with suspected CAD and stable angina symptoms and/or dyspnea; patients with new onset of heart failure or left ventricular dysfunction and suspected CAD; asymptomatic and symptomatic patients with stabilized symptoms within one year after an acute coronary syndrome, or patients with recent revascularisation; asymptomatic and symptomatic patients beyond one year after initial diagnosis or revascularisation; Patients with angina and suspected vasospastic or microvascular disease; Asymptomatic subjects in whom CAD is detected at screening. Although these scenarios are heterogeneous, they are associated with an increased risk of acute events, and the stability of CCS patients over time depends on prompt diagnosis, optimal treatment and secondary prevention strategies, including Lifestyle modifications, and pharmacotherapy.

ELIGIBILITY:
Inclusion criteria

Adult patients (18 years or older) with a confirmed or suspected diagnosis of CCS, fall within one of the following broad CCS categories:

* Patients with angina and/or dyspnea, and suspected coronary artery disease.
* Patients with new onset of heart failure or reduced left ventricular function.
* Patients within 1 year after an acute coronary syndrome or recent revascularization.
* Patients beyond 1 year after initial diagnosis or revascularization.
* Patients with ANOCA (e.g., microvascular angina, vasospastic angina).
* Asymptomatic subjects referred for screening for coronary artery disease.

Exclusion Criteria:

* Patients with a recent acute coronary syndrome (defined as those within 1 month of a diagnosis of unstable angina, non-ST-segment elevation myocardial infarction or ST-segment elevation myocardial infarction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with angina and/or dyspnea, and suspected coronary artery disease. Patients with new onset of heart failure or reduced left ventricular function. Patients within 1 year after an acute coronary syndrome or recent revascularization.
  Patients beyond 1 year after initial diagnosis or revascularization. Patients with ANOCA (e.g., microvascular angina, vasospastic angina). Asymptomatic subjects referred for screening for coronary artery disease.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-10-22 (Estimated); Study Completion 2025-10-22 (Estimated)

PRIMARY OUTCOMES:
effect of revasculariztion strategies on chronic coronary syndrome patients | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Department Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No